CLINICAL TRIAL: NCT04031833
Title: Encochleated Oral Amphotericin for Cryptococcal Meningitis Trial
Brief Title: Encochleated Oral Amphotericin for Cryptococcal Meningitis Trial (EnACT)
Acronym: EnACT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-70007
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B

STUDY DESIGN:
Intervention Model Description: Phase I: Persons in Uganda without meningitis or active infections Phase II: HIV-infected persons in Uganda with cryptococcal meningitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a single ascending dose study (Experimental): Phase IA will consist of a single ascending dose study in 9 participants to test three doses to determine the max tolerated dose.
  Interventions: Drug: MAT2203
- Phase 1b multiple day dosing (Experimental): 9 subjects will receive the Phase Ia 100% tolerated MAT2203 dose for 7 days.
  Interventions: Drug: MAT2203
- Phase 2 safety and tolerability (Experimental): Safety, tolerability, and microbiologic efficacy of MAT2203 among HIV-infected patients with cryptococcal meningitis compared with standard IV AMB.
  Interventions: Drug: MAT2203; Drug: Amphotericin B

INTERVENTIONS:
Drug: MAT2203 — Encochleated amphotericin B
  Other Names: oral amphotericin B
Drug: Amphotericin B — Intravenous amphotericin B
  Arms: Phase 2 safety and tolerability

SUMMARY:
This study is designed as two sequential trials. The first is a phase I open label trial to evaluate the safety and tolerability of MAT2203. The maximal tolerated and non-toxic daily dose,will then be moved forward into a multi-day safety trial. The Phase II trial will investigate toxicity and early fungicidal activity (EFA) of MAT2203 with flucytosine.

DETAILED DESCRIPTION:
Cryptococcal meningitis has emerged as one of the most frequent and deadly opportunistic infections in HIV patients. Historically, amphotericin B (AMB) has been considered the "gold standard" in antifungal treatments due to its broad spectrum of activity and lack of emergence of resistance. However, the use of AMB is limited by side effects, including nephrotoxicity, anemia, and infusion-related reactions. MAT2203 or encochleated oral amphotericin B (cAMB) is a lipid nano-crystal formulation designed for targeted oral delivery of the antifungal drug AMB for treatment of fungal and parasitic infections.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1:

  * Age >18 years
  * Calculated creatinine clearance >70 mL/min/1.73 m2 (measured within 3 months)
  * Written informed consent

Phase 2:

* Cryptococcal meningitis diagnosed by CSF cryptococcal antigen (CRAG)
* Ability and willingness to provide informed consent
* Willing to receive protocol-specified lumbar punctures

Exclusion Criteria:

* Phase 1:

  * Symptomatic Current illness
  * Known significant, untreated health problem
  * Inability to take enteral medicine
  * Pregnant or breast feeding
  * Receiving amphotericin B therapy in past 90 days
* Phase 2:

  * Presenting Glasgow Coma Scale (GCS) < 15
  * Received 3 or more doses of IV amphotericin therapy within last 30 days
  * Inability to take enteral (oral or nasogastric) medicine
  * Cannot or unlikely to attend regular clinic visits
  * Pregnancy or breastfeeding
  * Receiving chemotherapy or corticosteroids
  * Suspected Paradoxical immune reconstitution inflammatory syndrome (IRIS)
  * Recent initiation of HIV therapy or ART class switch (within 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Highest dose tolerated without inducing vomiting | 7 days
  Proportion of cAMB daily dose received and tolerated without vomiting within 30 minutes.
Evidence of fungicidal activity | 2 weeks
  CSF early fungicidal activity (EFA) during 2-week induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahimbisibwe C, Kwizera R, Ndyetukira JF, Namujju OC, Sadiq A, Atukunda M, Skipper CP, Boulware DR, Meya DB. Experience of research nurses with oral encochleated amphotericin B for treatment of cryptococcal meningitis in a resource-limited setting. BMC Infect Dis. 2025 Jul 15;25(1):920. doi: 10.1186/s12879-025-11319-1. PMID 40665233
- [Derived] Sadiq A, Kwizera R, Kiiza TK, Ayebare P, Ahimbisibwe C, Ndyetukira JF, Boulware DR, Meya DB. Experiences, challenges, gaps, and strategies for counselling persons presenting with advanced HIV-associated meningitis in Uganda. AIDS Res Ther. 2025 Feb 19;22(1):21. doi: 10.1186/s12981-025-00705-z. PMID 39972326
- [Derived] Kimuda S, Kwizera R, Dai B, Kigozi E, Kasozi D, Rutakingirwa MK, Tukundane A, Shifah N, Luggya T, Luswata A, Ndyetukira JF, Yueh SL, Mulwana S, Wele A, Bahr NC, Meya DB, Boulware DR, Skipper CP. Comparison of Early Fungicidal Activity and Mortality Between Daily Liposomal Amphotericin B and Daily Amphotericin B Deoxycholate for Cryptococcal Meningitis. Clin Infect Dis. 2025 Feb 5;80(1):153-159. doi: 10.1093/cid/ciae326. PMID 38943665
- [Derived] Boulware DR, Atukunda M, Kagimu E, Musubire AK, Akampurira A, Tugume L, Ssebambulidde K, Kasibante J, Nsangi L, Mugabi T, Gakuru J, Kimuda S, Kasozi D, Namombwe S, Turyasingura I, Rutakingirwa MK, Mpoza E, Kigozi E, Muzoora C, Ellis J, Skipper CP, Matkovits T, Williamson PR, Williams DA, Fieberg A, Hullsiek KH, Abassi M, Dai B, Meya DB. Oral Lipid Nanocrystal Amphotericin B for Cryptococcal Meningitis: A Randomized Clinical Trial. Clin Infect Dis. 2023 Dec 15;77(12):1659-1667. doi: 10.1093/cid/ciad440. PMID 37606364
- [Derived] Skipper CP, Atukunda M, Stadelman A, Engen NW, Bangdiwala AS, Hullsiek KH, Abassi M, Rhein J, Nicol MR, Laker E, Williams DA, Mannino R, Matkovits T, Meya DB, Boulware DR. Phase I EnACT Trial of the Safety and Tolerability of a Novel Oral Formulation of Amphotericin B. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e00838-20. doi: 10.1128/AAC.00838-20. Print 2020 Sep 21. PMID 32747357